CLINICAL TRIAL: NCT04591509
Title: Predictive Value of Diaphragmatic Excursion by Echographic Assessment at the Bedside on Need for Endotracheal Intubation in COPD Patients With Acute Dyspnea in Emergency Medicine
Brief Title: Predictability of Echographic Excursion of the Diaphragm for Intubation in COPD- Patients With Acute Respiratory Failure in ED
Acronym: PREEDICT-ED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Matthieu Daniel, Head of Clinic - Intensive Care Unit, European Georges Pompidou Hospital
Other Study IDs: EuroeanGPH
Record Dates: First submitted 2020-10-03; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: COPD Exacerbation; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators seek to evaluate if the ultra-sound measure of the diaphragm expansion is predictive of admission into an ICU and/or intubation for patients with COPD.

Every patient coming to the ER with shortness of breath and a known or suspected COPD, will undergo standard of care associated with a diaphragm ultrasound.

The investigators will then gather, through the internal databases of the recruiting hospitals, information about admission into ICU and/or intubation.

The investigators think that this technique will help improve early detection of COPD patient requiring mechanical ventilation, using ultrasound, a non invasive technique.

DETAILED DESCRIPTION:
Inclusion of every lawful age patient presenting to the ER with inclusion criterias

The patient must not have exclusion criteria and must have received the information and consent sheets to be signed jointly

Then, the investigators perform an online randomization for the first and second operator and the side (left/right) from which they start the ultrasound assessment.

The investigators then assess diaphragmatic excursion measurements in spontaneously ventilated patient at 45 ° proclive position for each hemi-diaphragm, with the 2 operators blinded to each other, for 3 consecutive respiratory cycles and save the images.

The date of inclusion is then reported in the register.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous ventilation at arrival to the ER
* With Respiratory Failure defined by at least of the following criterias :

  * Respiratory frequency > 25 and/or clinical signs of respiratory failure
  * Hypoxia with a WpO2 < 90%
  * Hypercapnia > 45mmHg with a respiratory acidosis

Exclusion Criteria:

* Known diaphragmatic dysfunction
* Necessity of immediate intubation leaving no time for ultrasound measurements of diaphragmatic excursion
* Unable to provide informed consent
* Evolutive or degenerative neurological disease that could affect diaphragmatic function
* Intracranial Hypertension
* Haemodynamic instability
* Acute heart failure
* Pregnant or Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient over 18, with known or suspected COPD, admitted to the ER for Respiratory Failure.
Sampling Method: Probability Sample
Enrollment: 390 (Estimated)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-01-23 (Estimated); Study Completion 2022-07-23 (Estimated)

PRIMARY OUTCOMES:
Evaluate the predictive value of the presence of diaphragmatic dysfunction diagnosed by ultrasound measurement of the diaphragmatic excursion (ED) on the use of invasive mechanical ventilation (IV) | During the 24 first hours after admission to the ED
  predictive value of the presence of a diaphragmatic dysfunction on the use of invasive mechanical ventilation (IV)

SECONDARY OUTCOMES:
Evaluate the predictive value of the ultrasound measurement of the E-T index for the use of invasive ventilation E-T index (IET) on the use of mechanical ventilation invasive | During the first 24 hours after admission to ED
  the E-T index for the use of invasive ventilation
Find a correlation between length of stay, length of ventilation, respiratory complications and the values of ED and E-T index measured at patient admission | Through study completion, an average of 2 years
  Duration of stay, ventilation (invasive and non-invasive), respiratory complications and the values of ED and E-T index
Assessment of staff learning curves senior and junior medical staff participating in initial training. | Through study completion, an average of 2 years
  Evaluation of learning curves
Assess the inter-observer feasibility and reproducibility of the measurement of ED and IET measured by ultrasound in time-movement mode (TM) | Through study completion, an average of 2 years
  Inter-operator feasibility and reproducibility of ED and IET

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu DANIEL, MD, Principal Investigator — European Georges Pompidou Hospital
Locations (3):
- France (3):
  - Nîmes University Hospital, Nîmes
  - Georges Pompidou European Hospital, Paris
  - Bellepierre Hospital, Saint-Denis

REFERENCES:
- [Background] Osadnik CR, Tee VS, Carson-Chahhoud KV, Picot J, Wedzicha JA, Smith BJ. Non-invasive ventilation for the management of acute hypercapnic respiratory failure due to exacerbation of chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2017 Jul 13;7(7):CD004104. doi: 10.1002/14651858.CD004104.pub4. PMID 28702957
- [Background] Guttikonda SNR, Vadapalli K. Approach to undifferentiated dyspnea in emergency department: aids in rapid clinical decision-making. Int J Emerg Med. 2018 Apr 4;11(1):21. doi: 10.1186/s12245-018-0181-z. PMID 29619581
- [Background] Palkar A, Narasimhan M, Greenberg H, Singh K, Koenig S, Mayo P, Gottesman E. Diaphragm Excursion-Time Index: A New Parameter Using Ultrasonography to Predict Extubation Outcome. Chest. 2018 May;153(5):1213-1220. doi: 10.1016/j.chest.2018.01.007. Epub 2018 Jan 17. PMID 29353023
- [Background] Bobbia X, Clement A, Claret PG, Bastide S, Alonso S, Wagner P, Tison T, Muller L, de La Coussaye JE. Diaphragmatic excursion measurement in emergency patients with acute dyspnea: toward a new diagnostic tool? Am J Emerg Med. 2016 Aug;34(8):1653-7. doi: 10.1016/j.ajem.2016.05.055. Epub 2016 May 24. PMID 27251231
- [Background] Boussuges A, Gole Y, Blanc P. Diaphragmatic motion studied by m-mode ultrasonography: methods, reproducibility, and normal values. Chest. 2009 Feb;135(2):391-400. doi: 10.1378/chest.08-1541. Epub 2008 Nov 18. PMID 19017880
- [Background] Marchioni A, Castaniere I, Tonelli R, Fantini R, Fontana M, Tabbi L, Viani A, Giaroni F, Ruggieri V, Cerri S, Clini E. Ultrasound-assessed diaphragmatic impairment is a predictor of outcomes in patients with acute exacerbation of chronic obstructive pulmonary disease undergoing noninvasive ventilation. Crit Care. 2018 Apr 27;22(1):109. doi: 10.1186/s13054-018-2033-x. PMID 29703214
- [Background] Zanobetti M, Scorpiniti M, Gigli C, Nazerian P, Vanni S, Innocenti F, Stefanone VT, Savinelli C, Coppa A, Bigiarini S, Caldi F, Tassinari I, Conti A, Grifoni S, Pini R. Point-of-Care Ultrasonography for Evaluation of Acute Dyspnea in the ED. Chest. 2017 Jun;151(6):1295-1301. doi: 10.1016/j.chest.2017.02.003. Epub 2017 Feb 16. PMID 28212836
- [Background] Malas O, Caglayan B, Fidan A, Ocal Z, Ozdogan S, Torun E. Cardiac or pulmonary dyspnea in patients admitted to the emergency department. Respir Med. 2003 Dec;97(12):1277-81. doi: 10.1016/j.rmed.2003.07.002. PMID 14682407
- [Background] Mueller C, Scholer A, Laule-Kilian K, Martina B, Schindler C, Buser P, Pfisterer M, Perruchoud AP. Use of B-type natriuretic peptide in the evaluation and management of acute dyspnea. N Engl J Med. 2004 Feb 12;350(7):647-54. doi: 10.1056/NEJMoa031681. PMID 14960741
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Rodriguez-Roisin R. Toward a consensus definition for COPD exacerbations. Chest. 2000 May;117(5 Suppl 2):398S-401S. doi: 10.1378/chest.117.5_suppl_2.398s. PMID 10843984
- [Background] Brochard L, Mancebo J, Wysocki M, Lofaso F, Conti G, Rauss A, Simonneau G, Benito S, Gasparetto A, Lemaire F, et al. Noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 1995 Sep 28;333(13):817-22. doi: 10.1056/NEJM199509283331301. PMID 7651472
- [Background] Bobbia X, Hansel N, Muller L, Claret PG, Moreau A, Genre Grandpierre R, Chenaitia H, Lefrant JY, de La Coussaye JE. Availability and practice of bedside ultrasonography in emergency rooms and prehospital setting: a French survey. Ann Fr Anesth Reanim. 2014 Mar;33(3):e29-33. doi: 10.1016/j.annfar.2013.12.010. Epub 2014 Jan 20. PMID 24456614
- [Background] Antenora F, Fantini R, Iattoni A, Castaniere I, Sdanganelli A, Livrieri F, Tonelli R, Zona S, Monelli M, Clini EM, Marchioni A. Prevalence and outcomes of diaphragmatic dysfunction assessed by ultrasound technology during acute exacerbation of COPD: A pilot study. Respirology. 2017 Feb;22(2):338-344. doi: 10.1111/resp.12916. Epub 2016 Oct 14. PMID 27743430
- [Background] De Troyer A, Wilson TA. Effect of acute inflation on the mechanics of the inspiratory muscles. J Appl Physiol (1985). 2009 Jul;107(1):315-23. doi: 10.1152/japplphysiol.91472.2008. Epub 2009 Mar 5. PMID 19265064
- [Background] Gayan-Ramirez G, Decramer M. Mechanisms of striated muscle dysfunction during acute exacerbations of COPD. J Appl Physiol (1985). 2013 May;114(9):1291-9. doi: 10.1152/japplphysiol.00847.2012. Epub 2013 Jan 31. PMID 23372146
- [Background] Unal O, Arslan H, Uzun K, Ozbay B, Sakarya ME. Evaluation of diaphragmatic movement with MR fluoroscopy in chronic obstructive pulmonary disease. Clin Imaging. 2000 Nov-Dec;24(6):347-50. doi: 10.1016/s0899-7071(00)00245-x. PMID 11368935
- [Background] Doucet M, Debigare R, Joanisse DR, Cote C, Leblanc P, Gregoire J, Deslauriers J, Vaillancourt R, Maltais F. Adaptation of the diaphragm and the vastus lateralis in mild-to-moderate COPD. Eur Respir J. 2004 Dec;24(6):971-9. doi: 10.1183/09031936.04.00020204. PMID 15572541
- [Background] Demoule A, Girou E, Richard JC, Taille S, Brochard L. Benefits and risks of success or failure of noninvasive ventilation. Intensive Care Med. 2006 Nov;32(11):1756-65. doi: 10.1007/s00134-006-0324-1. Epub 2006 Sep 21. PMID 17019559
- [Background] Levine S, Nguyen T, Kaiser LR, Rubinstein NA, Maislin G, Gregory C, Rome LC, Dudley GA, Sieck GC, Shrager JB. Human diaphragm remodeling associated with chronic obstructive pulmonary disease: clinical implications. Am J Respir Crit Care Med. 2003 Sep 15;168(6):706-13. doi: 10.1164/rccm.200209-1070OC. Epub 2003 Jul 11. PMID 12857719
- [Background] Levine S, Kaiser L, Leferovich J, Tikunov B. Cellular adaptations in the diaphragm in chronic obstructive pulmonary disease. N Engl J Med. 1997 Dec 18;337(25):1799-806. doi: 10.1056/NEJM199712183372503. PMID 9400036
- [Background] Sinderby C, Spahija J, Beck J, Kaminski D, Yan S, Comtois N, Sliwinski P. Diaphragm activation during exercise in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2001 Jun;163(7):1637-41. doi: 10.1164/ajrccm.163.7.2007033. PMID 11401887
- [Background] Hughes PD, Polkey MI, Harrus ML, Coats AJ, Moxham J, Green M. Diaphragm strength in chronic heart failure. Am J Respir Crit Care Med. 1999 Aug;160(2):529-34. doi: 10.1164/ajrccm.160.2.9810081. PMID 10430724
- [Background] Watson RA, Pride NB. Postural changes in lung volumes and respiratory resistance in subjects with obesity. J Appl Physiol (1985). 2005 Feb;98(2):512-7. doi: 10.1152/japplphysiol.00430.2004. Epub 2004 Oct 8. PMID 15475605
- [Background] McCool FD, Tzelepis GE. Dysfunction of the diaphragm. N Engl J Med. 2012 Mar 8;366(10):932-42. doi: 10.1056/NEJMra1007236. No abstract available. PMID 22397655
- [Derived] Markarian T, Daniel M, Guillemet K, Ajavon F, Femy F, Grandpierre RG, Feral-Pierssens AL, Bobbia X. Visual Patterns of Diaphragmatic Motion in Acute Respiratory Failure: A Prospective Pilot Study. J Clin Ultrasound. 2025 Mar-Apr;53(3):421-428. doi: 10.1002/jcu.23886. Epub 2024 Oct 29. PMID 39470416